CLINICAL TRIAL: NCT05790213
Title: Phase II Trial of Focal Prostate Ablation Combined With Androgen Deprivation Therapy for Prostate Cancer Treatment
Brief Title: Prostate Cancer Treatment Using Androgen Deprivation Therapy and Focal Prostate Ablation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0259
Record Dates: First submitted 2023-02-07; First posted 2023-03-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive Androgen deprivation therapy (ADT) followed by Focal prostate ablation (focal therapy)
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Procedure: Focal prostate ablation (focal therapy)

INTERVENTIONS:
Drug: Androgen Deprivation Therapy (ADT) — ADT will be given for 3 months. Participants will receive a standard ADT as chosen by their study doctor.
Procedure: Focal prostate ablation (focal therapy) — Focal prostate ablation (focal therapy) is a surgical procedure to destroy cancer cells by destroying a portion of the prostate instead of the whole prostate.

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of combining focal prostate ablation therapy ((aka Focal Therapy, a surgical procedure) and androgen deprivation therapy (hormone therapy).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have intermediate-risk PCa as defined by the below criteria:

  a. Favorable intermediate-risk PCa: i. ≤ clinical stage T2c, GG2, and PSA ≤ 10 ng/mL, and <50% positive biopsy cores with PCa b. Unfavorable intermediate-risk PCa: i. ≤ clinical stageT2c, GG2, and PSA 10-20 ng/mL, or ≥50% positive biopsy cores with PCa, or ii. ≤ clinical stage T2c, GG3, and PSA < 20 ng/mL
* No mpMRI evidence of extra-prostatic extension (EPE) or seminal vesicle invasion, and if seminal vesical invasion is suspected, it must be excluded by prostate biopsy.
* Subjects must have chosen to get Focal Therapy for the treatment of prostate cancer.
* Subjects must have confirmed non-metastatic PCa following SOC screening for patients with unfavorable intermediate-risk PCa, a combination of computed tomography imaging of the abdomen and pelvis (CTAP) and technetium-99-mDP nuclear medicine bone scan (BS) and/or prostate-specific membrane antigen positron emission tomography (PSMA/PET) scan prior to enrollment. The imaging studies should be obtained within 6-months of enrollment. Additional imaging is not required for men with favorable intermediate-risk PCa.
* Subject must be male ≥ 18 years-old.
* Subjects must have a life expectancy of at least 10-years per the opinion of the treating investigator.
* Subjects must be designated as Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky Performance Status Scale Score ≥ 60%, see Appendix A).
* Subjects must be fit to undergo general anesthesia and the FT surgical procedure, which includes adequate visualization of the prostate gland on transrectal ultrasound imaging, access to the urethra, perineum and rectum, as well as be tolerant of lithotomy positioning in the opinion of the treating investigator or the operating surgeon(s) if not the same as the treating investigator.
* Subjects must have adequate organ and marrow function as defined below:

Hemoglobin ≥ 10 g/dL Leukocytes ≥ 3,000/mcL Absolute neutrophil count ≥ 1,500/mcL Platelets ≥ 100,000/mcL Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN Creatinine < 1.5 institutional ULN OR Calculated or measured creatinine clearance > 50 mL/min/1.73 m2 eGFR >30 mL/min using the MDRD (modification of diet and renal disease) formula Serum albumin ≥3.0 g/dL Serum potassium ≥3.5 mmol/L

* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Subjects who are sexually active with a woman of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and his partner must also be practicing a highly effective method of contraception (i.e., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system) during treatment and for 3-months following the last ADT treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subject has had prior or current PCa therapies, such as biologic, chemotherapy, hormone therapy, radiotherapy or surgery for PCa. Subjects may not have had undergone pelvic radiation, chemotherapy or immunotherapy treatment for a separate hematologic or visceral malignancy within 6-months of enrollment in the present study.
* Subjects with locally advanced, nodal or metastatic prostate cancer.
* Subjects who are unfit for pelvic mpMRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, metallic implants that are likely to contribute to significant image artifacts, allergy or contraindication to gadolinium contrast agent.
* History of allergy or intolerance to study drug components.
* History of bilateral orchiectomy.
* If the subject has an uncontrolled or major debilitating inter-current illness.
* Subjects who are receiving any other investigational agents, or who have received other investigational agents in the past and who are no longer receiving these investigational agents may be eligible at the discretion of the principal investigator (PI).
* Judgment by the treating investigator or PI that the subject is unsuitable to participate in the study and the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 57 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-12-18 (Estimated); Study Completion 2028-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinically significant residual prostate cancer in ablated prostate tissue following study treatment | End of Treatment (approximately 4-5 months)
  Proportion of participants that have residual cancer in ablated prostate tissue. Residual disease will be measured by MRI.
Number of participants with clinically significant residual prostate cancer in unablated prostate tissue following study treatment | End of Treatment (approximately 4-5 months)
  Proportion of participants that have residual cancer in unablated prostate tissue. Residual disease will be measured by MRI.
Number and grade of complications [Safety] | 6-months following treatment
  Number and grade of complications will be reported.
  Number and grade of complications will be reported.
  The number and severity by Common Terminology Criteria for Adverse Events (CTCAE) grade of reported complications will be reported.

SECONDARY OUTCOMES:
Measuring change in genitourinary and sexual function and health-related quality of life (measured by HRQoL) | 6-and 12-months after FT
  Define change in genitourinary and sexual function from baseline following ADT and FT by measuring the subject's HRQoL
PSA response to the combination treatment | Baseline, 3-months, 6-months, and 1-year from FT
  Determine the PSA response to the combination treatment by measuring the subject's PSA at "baseline" (PSA at time of initial diagnosis) 3-months, 6-months, and 1-year from FT
Proportion of men converting therapy or dying of prostate cancer during study | 12 months after FT
  Determine the proportion of men converting to whole gland therapy (radical prostatectomy or radiation therapy) and/or requiring systemic therapy and/or developing metastases and/or dying of PCa during the course of study.
Post Treatment biopsy with no prostate cancer | 6 months after FT
  Determine the proportion of men without any prostate cancer on any post treatment prostate biopsy.
Proportion of men with normal baseline serum | 6-, 9- and 12-months after FT.
  Determine the proportion of men with normal baseline serum testosterone who had testosterone recovery (defined as testosterone levels >300 ng/dL) at 6-, 9- and 12-months after FT.
  Testosterone recovery: Number of men who have recovered normal serum testosterone levels will be expressed as proportions of total number of eugonadal patients and the 95% confidence interval of the proportion will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sidana, MD, Principal Investigator — University of Chicago
Locations (1):
- UChicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koehler J, Lama D, Mendez M, Hsu WW, Oto A, Szmulewitz R, Sidana A. Phase II trial protocol of focal prostate ablation combined with androgen deprivation therapy for prostate cancer treatment. PLoS One. 2025 Dec 16;20(12):e0337828. doi: 10.1371/journal.pone.0337828. eCollection 2025. PMID 41401176